CLINICAL TRIAL: NCT03760419
Title: Improving CarE for Community Acquired Pneumonia 1 (ICE-CAP1): Antibiotic Decision Support
Brief Title: Improving CarE for Community Acquired Pneumonia 1
Acronym: ICE-CAP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Derek Williams, Derek Williams, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AI125642 (NIH); R01AI125642 (NIH)
Record Dates: First submitted 2018-09-15; First posted 2018-11-30 (Actual); Results first posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Pneumonia Childhood

STUDY DESIGN:
Intervention Model Description: Effectiveness of the EHR-based antibiotic decision support application for promoting guideline-concordant antibiotic prescribing in children presenting for emergency care will be evaluated in a pragmatic, cluster-randomized study conducted over a period of 18 months that includes two respiratory seasons. Randomization will occur monthly at each hospital. To ensure balanced representation of each arm in periods of both low and high pneumonia prevalence, randomization will occur in 3 permuted blocks (size=6).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The antibiotic decision support application will be provided to those randomized to the intervention arm. Due to the nature of the intervention, blinding of treating providers will not be possible. All children will receive usual care and all treatment decisions will be made by the clinical providers and will not be restricted or altered in any way.
  Interventions: Behavioral: Clinical Decision Support
- Control Arm (No Intervention): No experimental decision support will be provided to those randomized to the control arm. All children will receive usual care and treatment will not be restricted or altered in any way by the study.

INTERVENTIONS:
Behavioral: Clinical Decision Support — For enrolled subjects assigned to the decision support arm, providers will receive antibiotic recommendations in accordance with the 2011 PIDS/IDSA guideline, tailored to site of care and illness severity. The tool will offer treatment recommendations only and will not proscribe a specific treatment plan.
  Arms: Intervention Arm

SUMMARY:
Children with pneumonia presenting to the emergency department at Monroe Carell Jr. Children's Hospital at Vanderbilt or Children's Hospital of Pittsburgh will be potentially eligible for study. During intervention periods, providers caring for enrolled children will be presented with a detailed decision support strategy that emphasizes management in accordance with national guideline recommendations. The anticipated study duration is 18 months and, as this study does not include direct contact with enrolled subjects, there is no anticipated follow up.

DETAILED DESCRIPTION:
Pneumonia is the most common serious infection in childhood. In the United States (US), pneumonia accounts for 1-4% of all emergency department (ED) visits in children (3-28 per 1,000 US children per year) and ranks among the top 3 reasons for pediatric hospitalization with >100,000 hospitalizations per year (15-22 per 100,000 US children per year)2-5. Pneumonia also accounts for more days of antibiotic use in US children's hospitals than any other condition.

Safely reducing inappropriate antibiotic use is critical to slow the progression of antimicrobial resistance, and childhood pneumonia is a key area where substantial improvements can be made. In the 2011 Pediatric Infectious Diseases Society/Infectious Diseases Society of America (PIDS/IDSA) pneumonia guideline, appropriate use of antibiotics was an important area of emphasis. For presumed bacterial pneumonia, recommendations emphasize the use of a single, narrow-spectrum antibiotic (i.e. amoxicillin or ampicillin). In children <6 years of age treated in the outpatient setting, the guideline recommended considering withholding antibiotics, recognizing that pneumonia in this population is most often caused by viruses. Both of these recommendations were graded as strong and supported by high-quality evidence. Nonetheless, in a large database study we conducted just prior to release of the 2011 guideline, use of broad-spectrum antibiotics was very common among children hospitalized with pneumonia, with substantial differences in antibiotic selection patterns among the various hospitals. In that study, use of narrow-spectrum ampicillin was rare (<5%). High rates of broad-spectrum antibiotic use were also noted in a study of children with pneumonia treated and released from US EDs, with <30% of children receiving narrow-spectrum therapy.

Study Aim: To test the hypothesis that electronic antibiotic decision support increases guideline-concordant antibiotic use compared with usual care in the emergency department.

The primary outcome is the proportion of children exclusively receiving guideline-concordant first line antibiotic therapy during the first 24 hours of care. Secondary outcomes include exclusive use of concordant antibiotic therapy for the entire episode, any use of concordant antibiotic therapy during the first 24 hours of care and for the entire episode, and emergency department revisits and hospitalizations within 72 hours and 7 days of the index discharge.

In this study, conducted at two experienced academic centers, the investigator will implement and evaluate an electronic health record based clinical decision support application to promote antibiotic use in concordance with the 2011 PIDS/IDSA guideline in a pragmatic, cluster randomized trial. Decisions regarding management, including antibiotic selection and site of care, will be at the discretion of the treating provider and will not be restricted or altered in any way. Thus, this study poses no greater than minimal risks to participants. Due to the nature of the research, waiver of informed consent has been provided, as it has been done in similar pragmatic studies at the institutions.

ELIGIBILITY:
Inclusion Criteria:

* Six months to <18 years of age
* Radiographic evidence of pneumonia in ED
* Provider-confirmed diagnosis of pneumonia (via Clinical Decision Support [CDS])

Exclusion Criteria:

* Children with tracheostomy, cystic fibrosis, immunosuppression
* Inter-hospital transfers
* Hospitalization within preceding 7 days
* Previously enrolled within preceding 28 days
* Provider preference for any reason

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1027 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Williams, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital - Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Monroe Carell Jr Children's Hospital at Vanderbilt; Children's Hospital of Pittsburgh: Children with pneumonia presenting to the ED at Monroe Carell Jr. Children's Hospital at Vanderbilt. Encounters were randomized to control or intervention.
  Control: Standard of care will be provided to those randomized to the control arm.
  Intervention: The antibiotic decision support application will be provided to those randomized to the intervention arm.
Period: Overall Study
Arm/Group | Monroe Carell Jr Children's Hospital at Vanderbilt | Children's Hospital of Pittsburgh
Started | 535 | 492
Received Intervention | 214 | 335
Received Contol | 321 | 157
Completed | 535 | 492
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention Arm | Total
Number analyzed (Participants) | 478 | 549 | 1027
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.8 [2.2 to 9.5] | 4.0 [1.7 to 7.4] | 4.2 [1.9 to 8.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 246 | 463
  Male | 261 | 303 | 564
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 36 | 96
  Not Hispanic or Latino | 390 | 472 | 862
  Unknown or Not Reported | 28 | 41 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 294 | 399 | 693
  Black | 117 | 79 | 196
  Asian | 14 | 17 | 31
  Mixed | 10 | 12 | 22
  Other | 24 | 20 | 44
  Unknown | 19 | 22 | 41
Comorbidity [Count of Participants; unit: Participants]
  Non-Chronic | 282 | 359 | 641
  Non-complex Chronic | 61 | 70 | 131
  Complex Chronic | 135 | 120 | 255
Insurance [Count of Participants; unit: Participants] — Population: This measurement was not able to be assessed for 3 patients.
  Participants
    number analyzed (Participants) | 475 | 549 | 1024
    Public | 281 | 280 | 561
    Private | 176 | 246 | 422
    Self-Pay | 18 | 23 | 41
Temperature [Median (Inter-Quartile Range); unit: degrees Celsius] | 37.3 [36.8 to 38.1] | 37.5 [36.9 to 38.4] | 37.4 [36.9 to 38.3]
Heart rate [Median (Inter-Quartile Range); unit: bpm] | 134 [113 to 153] | 139 [120 to 159] | 136 [116 to 156]
Respiratory rate [Median (Inter-Quartile Range); unit: respirations per minute] — BPM (breaths/min)
  respirations per minute | 30 [24 to 40] | 34 [24 to 46] | 32 [24 to 44]
Systolic BP [Median (Inter-Quartile Range); unit: mmHg] | 108 [100 to 117] | 108 [100 to 116] | 108 [100 to 116]
SpO2:FiO2 ratio [Median (Inter-Quartile Range); unit: ratio] | 462 [360 to 479] | 457 [306 to 474] | 457 [328 to 474]
ED Disposition [Count of Participants; unit: Participants]
  Home | 212 | 219 | 431
  Inpatient | 189 | 215 | 404
  Intensive Care | 77 | 115 | 192
Enrolling Site [Count of Participants; unit: Participants]
  Site A | 321 | 214 | 535
  Site B | 157 | 335 | 492

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Guideline-Concordant Antibiotic Therapy, First 24 Hours
Description: The primary outcome is the percentage of children in which ALL antibiotic treatment prescribed in the first 24 hours of the encounter is guideline-concordant.
Time Frame: 18 months
Population: All categories except "Overall" are subsets of the overall number. The category for each row shows the percentage of that subset that meets the specific criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 478 | 549
Participants
  Overall | 255 | 284
  Site A: number analyzed (Participants) | 321 | 214
  Site A | 174 | 120
  Site B: number analyzed (Participants) | 157 | 335
  Site B | 81 | 164
  Outpatient: number analyzed (Participants) | 212 | 219
  Outpatient | 140 | 164
  Inpatient: number analyzed (Participants) | 189 | 215
  Inpatient | 93 | 99
  ICU: number analyzed (Participants) | 77 | 115
  ICU | 22 | 21
  Age < 6 years: number analyzed (Participants) | 280 | 359
  Age < 6 years | 163 | 192
  Age >/= 6 years: number analyzed (Participants) | 198 | 190
  Age >/= 6 years | 92 | 92
  Receiving Antibiotics: number analyzed (Participants) | 370 | 455
  Receiving Antibiotics | 147 | 192

2. Secondary Outcome: Exclusive Guideline-Concordant Antibiotic Prescribing, Entire Episode
Description: This secondary outcome reports encounters in which established antibiotic stewardship guidelines are followed for ALL prescribing for the duration of the encounter (ED triage through hospital discharge).
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 478 | 549
Participants
  Overall | 240 | 261
  Site A: number analyzed (Participants) | 321 | 214
  Site A | 163 | 111
  Site B: number analyzed (Participants) | 157 | 335
  Site B | 77 | 150
  Outpatient: number analyzed (Participants) | 212 | 219
  Outpatient | 140 | 164
  Inpatient: number analyzed (Participants) | 189 | 215
  Inpatient | 83 | 85
  ICU: number analyzed (Participants) | 77 | 115
  ICU | 17 | 12
  Age <6 years: number analyzed (Participants) | 280 | 359
  Age <6 years | 156 | 175
  Age >/= 6 years: number analyzed (Participants) | 198 | 190
  Age >/= 6 years | 84 | 86
  Receiving Antibiotics: number analyzed (Participants) | 373 | 462
  Receiving Antibiotics | 135 | 175

3. Secondary Outcome: Any Guideline-Concordant Antibiotic Prescribing, First 24 Hours
Description: This secondary outcome includes ANY guideline-concordant prescribing during the first 24 hours of the encounter.
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 478 | 549
Participants
  Overall | 297 | 358
  Site A: number analyzed (Participants) | 321 | 214
  Site A | 198 | 144
  Site B: number analyzed (Participants) | 157 | 335
  Site B | 99 | 214
  Outpatient: number analyzed (Participants) | 212 | 219
  Outpatient | 145 | 168
  Inpatient: number analyzed (Participants) | 189 | 215
  Inpatient | 117 | 145
  ICU: number analyzed (Participants) | 77 | 115
  ICU | 35 | 45
  Age <6 years: number analyzed (Participants) | 280 | 359
  Age <6 years | 189 | 242
  Age >/= 6 years: number analyzed (Participants) | 198 | 190
  Age >/= 6 years | 108 | 116
  Receiving Antibiotics: number analyzed (Participants) | 370 | 455
  Receiving Antibiotics | 189 | 266

4. Secondary Outcome: Any Guideline-Concordant Antibiotic Prescribing, Entire Episode
Description: This secondary outcome includes ANY guideline-concordant prescribing during the ENTIRE encounter (ED triage through hospital discharge).
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 478 | 549
Participants
  Overall | 305 | 383
  Site A: number analyzed (Participants) | 321 | 214
  Site A | 200 | 146
  Site B: number analyzed (Participants) | 157 | 335
  Site B | 105 | 237
  Outpatient: number analyzed (Participants) | 212 | 219
  Outpatient | 145 | 168
  Inpatient: number analyzed (Participants) | 189 | 215
  Inpatient | 119 | 154
  ICU: number analyzed (Participants) | 77 | 115
  ICU | 41 | 61
  Age <6 years: number analyzed (Participants) | 280 | 359
  Age <6 years | 195 | 256
  Age >/= 6 years: number analyzed (Participants) | 198 | 190
  Age >/= 6 years | 110 | 127
  Receiving Antibiotics: number analyzed (Participants) | 373 | 462
  Receiving Antibiotics | 200 | 297

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse event reporting will focus exclusively on ED revisits and/or inpatient hospital re-admissions within 3- or 7-days from index discharge and death within 30 days of index discharge. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | Control Arm | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 2/478 | 1/549
Serious Adverse Events (participants affected / at risk) | 83/478 | 74/549
Other Adverse Events (participants affected / at risk) | 0/478 | 0/549
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=478) | Intervention Arm (N=549)
ED revisit within 72 hours (Respiratory, thoracic and mediastinal disorders) | 19 | 22 — Patient returns to the Emergency Department within 72 hours for same illness as index visit.
ED revisit within 7 days (Respiratory, thoracic and mediastinal disorders) | 32 | 30 — Patient returns to the Emergency Department within 7 days for same illness as index visit.
Re-hospitalization within 72 hours (Respiratory, thoracic and mediastinal disorders) | 9 | 7 — Patient is admitted to the hospital within 72 hours for same illness as index visit.
Re-hospitalization within 7 days (Respiratory, thoracic and mediastinal disorders) | 23 | 15 — Patient is admitted to the hospital within 7 days for same illness as index visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03760419/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03760419/SAP_001.pdf